CLINICAL TRIAL: NCT06585761
Title: Effect of Sodium Glucose Co-tansporter 2 Inhibitors (SGLT2I) on Inflammatory and Oxidative Stress Markers Level in Heart Failure Patients
Status: Recruiting | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Nada Nabil Elsalhey, Dr, Kafrelsheikh University
Other Study IDs: KFSIRB200-128
Record Dates: First submitted 2024-08-23; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Sodium-Glucose Transporter 2 Inhibitors; empagliflozin; dapagliflozin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- pre-SGLT2I group: patients with heart failure newly introduced to one of SGLT2I members
  Interventions: Device: echo cardiogram
- Post-SGLT2I group: patients with heart failure on one of SGLT2I members for at least 2 months
  Interventions: Drug: SGLT2 inhibitor; Device: echo cardiogram

INTERVENTIONS:
Drug: SGLT2 inhibitor — patients with HF are subjected to regular dose of SGLT2I member according to patient status.
  Other Names: empagliflozin, Dapagliflozin
  Groups: Post-SGLT2I group
Device: echo cardiogram — the patients are subjected to ECHO to determine their EF prior to and post the study

SUMMARY:
The aim of this study is to explore the effect of SGLT2i on the levels of cardiac biomarkers, inflammatory and stress markers in Egyptian heart failure patients to provide a better understanding of mechanism that might assist in tailoring treatment strategies in patients with various forms of HF especially in Egyptian population. Also understand how biomarkers may be employed to predict risk in patients receiving SGLT2i or identification of those who may derive the most benefit from SGLT2i in the means of individualized medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged more than 18 years old.
2. Patients are with cardiac function was graded as II-IV by the New York Heart Association (NYHA)
3. Patients are on standard therapy for management of HF (according to AHA/ACC/HFSA Guideline for the Management of Heart Failure2022)21 such as:

   * ACEi (angiotensin converting enzyme inhibitor)
   * ARB (angiotensin receptor blocker)
   * ARNI in place of ACEi OR ARB
   * Beta blocker
   * (MRA) Mineralocorticoid receptor antagonists
   * Diuretics as needed.
4. All patients signed the informed consent.

Exclusion Criteria:

1. Patients suffering from conditions like acute CVS illness and severe sepsis that raise inflammatory markers and may lead to cardiac dysfunction as opposed to heart failure.
2. Patients with various cardiac conditions, such as severe congenital heart disease, myocarditis, and valvular heart disease.
3. Female patients during pregnancy or lactation
4. Individuals suffering from a malignant tumor, hyperfunctioning thyroid, multiple organ failure, or significantly reduced kidney function (eGFR <20 mL/min/1.73 m²).
5. Individuals suffering from verbal communication disorders or psychic cognitive impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants who are candidates for SGLT2i and will be recruited from Cardiology Department, Kafrelshiekh University Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
measure effect of SGLT2I ON serum concentration ( level) of cardiac biomarkers in heart failure patients before and after the intervention | 1 year
  At follow up, patients will be clinically evaluated for the changes in serum levels of the studied biomarkers the studied biomarker is NT-proBNP, its concentration is measured in pg/mL.
clinical examination for the presence and extent of improvement in signs and symptoms | 1 year
  Clinical examination depending on NYHA classification of the participants

SECONDARY OUTCOMES:
measure effect of SGLT2I ON serum concentration ( level) of cardiac inflammatory marker ( IL-6) in heart failure patients before and after the intervention | 1 year
  At follow up, patients will be clinically evaluated for the changes in serum levels of the studied biomarker
  Il-6 serum concentration is measured in pg/mL
Measure the effect of SGLT2I on serum concentration ( level) of cardiac inflammatory marker ( TNF-Alpha) in heart failure patients before and after the intervention | 1 year
  TNF-Alpha serum concentration is measured in pg/ml

OTHER OUTCOMES:
measure effect of SGLT2I ON serum concentration( level) of cardiac stress markers in heart failure patients before and after the intervention | 1 year
  At follow up, patients will be clinically evaluated for the changes in serum levels of the studied biomarkers such as MDA which plasma concentration is measured in nM

CONTACTS AND LOCATIONS:
Overall Officials: Nada Nabil Mohammed Elsalhey, Bsc, Principal Investigator — clinical pharmacy department, kafrelsheikh university
Locations (1):
- Kafrelsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided by participant